CLINICAL TRIAL: NCT04018534
Title: Effectiveness of Three Different Types Educational Methods on Implementation of Proper Oral Hygiene Behaviour Prior to Orthodontic Treatment
Brief Title: Effects Of Training On Brushing Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Fethiye Cakmak Ozlu (Unknown); Erol Aktunc (Unknown); Ersan Ilsay Karadeniz (Unknown)
Responsible Party: Principal Investigator, Hakan Yilmaz, Assistant Professor, Okan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11022014
Record Dates: First submitted 2019-07-07; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Orthodontic Appliances; Oral Health Training; Oral Hygiene

STUDY DESIGN:
Intervention Model Description: 90 consecutive fixed orthodontic appliance treatment candidates in compliance with the above mentioned criteria were randomly assigned to 3 groups (n = 30 in each); Control group: The patients in control group received a standard printed educational material assisted with verbal information in accordance with BOS educational goals.
  Study group 1: The patients in one of the study groups received a video assisted education .
  Study group 2: The patients in other study group received a hands-on training.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): The patients in control group received a standard printed educational material assisted with verbal information in accordance with British Orthodontics Society(BOS) educational goals.
  Interventions: Behavioral: Standard Verbal/Written Education
- Video assisted education group (Experimental): The patients in one of the study groups received a video assisted education
  Interventions: Behavioral: Video Assisted Education
- Hands-on training group (Experimental): The patients in other study group received a hands-on training.
  Interventions: Behavioral: Hands-on Training

INTERVENTIONS:
Behavioral: Standard Verbal/Written Education — This patients as control group received a standard printed educational material assisted with verbal information in accordance with British Orthodontics Society (BOS) educational goals.
  Arms: Control group
Behavioral: Video Assisted Education — The video training consisted of two separate sessions, each one lasting 5 minutes, one about the treatment materials and the other about the oral hygiene successively and in compliance with the British Orthodontics Society (BOS) educational obligations. All of the candidates were allowed to rewind and watch the video presentation until they reach all of the educational goals. The accomplishment of the educational goals was documented through a written examination form filled in by the candidates themselves. All of the candidates have rated fullscore in the written examinations on both topics.
  Arms: Video assisted education group
Behavioral: Hands-on Training — The hands-on training consisting of two separate sessions was performed by one of the authors (E.A). The first is about the treatment materials and the second one is about the oral hygiene successively. They are in accordance with the British Orthodontics Society (BOS) educational obligations. All of the patients were allowed to ask questions freely until they reach all of the educational goals. The accomplishments of the educational goals were documented through a written examination form filled in by the candidates themselves. All of the candidates have rated fullscore in the written examinations on both topics. The time requirements for all three different educational interventions were recorded separately.
  Arms: Hands-on training group

SUMMARY:
This study is a single-blind randomized controlled trial on fixed orthodontic appliance candidates (n = 90) assigned into a control group (n = 30) and two different study groups (n = 30 in each). Patients who requiring non-extraction fixed orthodontic treatment, crowding under 5mm in the incisors and heaving at least 20 permanent teeth with healthy periodontal tissue and devoid of caries were included in the study. The control group received a standard printed educational material assisted with verbal information. The study groups either received video assisted or hands-on training about fixed orthodontic appliance and oral hygiene. The time requirements for all three educational interventions were recorded at the initial visit. The adequacy of oral hygiene is documented through plaque and gingival indices at the initial visit and 8th week of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Required non-extraction fixed orthodontic treatment, agree to use conventional stainless steel brackets (Gemini series; 3M Unitek, Monrovia, California, USA), at least 20 natural permanent teeth, crowding under 5 mm in the incisors and willing to participate in our research

Exclusion Criteria:

* Dental caries, periodontal disease, systemic or chronic diseases such as diabetes, physical or mental disorders, smoking, previous orthodontic treatment, extensive dental restorations, antibiotic use during the previous 3 months, dental fluorosis and use of powered tooth brushes.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2018-11-24 (Actual)

PRIMARY OUTCOMES:
Plaque index(PI) for oral health assessment. | PI was measured at the 8 weeks later in each patient.
  The brushing habits of the patients were checked at each appointment and were recorded with PI. This measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth.
Gingival index(GI) for oral health assessment. | GI was measured at the 8 weeks later in each patient.
  This index was used to assess the severity and prevalence of gingivitis.Probe was used as a sensor for GI scoring and the mesial, distal, buccal and lingual surfaces of the teeth were evaluated in patients undergoing fixed orthodontic treatment.

SECONDARY OUTCOMES:
Time duration spent for educational interventions | Average 30 minutes
  The time requirements for all three different educational interventions were recorded separately.These time durations consisted of the education time needed for both fixed appliance components and oral hygiene educations all together.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozlu FC, Aktunc E, Yilmaz H, Karadeniz EI. Effectiveness of three different types of educational methods on implementation of proper oral hygiene behaviour prior to orthodontic treatment. Dental Press J Orthod. 2021 Mar 22;26(1):e2119248. doi: 10.1590/2177-6709.26.1.e2119248.oar. eCollection 2021. PMID 33759964